CLINICAL TRIAL: NCT02326038
Title: Can Methylphenidate (Ritalin) Improve Memory and Attention in Mild Cognitive Impairment? A Combined Behaviour-EEG Study
Brief Title: Ritalin, Memory and Attention in MCI: a Behaviour-EEG Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Orbis Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14T111; 2014-003117-28 (EudraCT Number)
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory; Attention; MCI; Ritalin
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ritalin (Experimental): Methylphenidate, capsule, 20 mg, single oral administration
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Placebo, capsule, single oral administration

INTERVENTIONS:
Drug: Methylphenidate — single oral administration of 20 mg tablet
  Other Names: Ritalin
  Arms: Ritalin

SUMMARY:
Traditionally, memory impairments in the elderly population are treated using cholinesterase inhibitors, although impairments remain after treatment. Dopamine (DA) is also involved in cognition and is especially of interest in healthy ageing because of the role in processing speed and cognitive control. To what extent dopamine treatment improves memory and attention in older impaired individuals is unknown. However, such an effect is conceivable because of the close relationship between memory and attention in aging and since improved processing speed and cognitive control may lead to improved memory.

The investigators aim to examine, in the impaired older population, whether a treatment using methylphenidate, a DA re-uptake inhibitor that enhances DA, improves attention and memory. The study will be conducted according to a cross-sectional, double-blind, placebo-controlled, 2-way cross-over design. 20 male and female patients with Mild Cognitive Impairment (MCI), amnestic type, aged above 60 years of age; 20 male and female patients with MCI, non-amnestic type, will be recruited from the Orbis Medical Centre. Participants will be treated once with 20 mg methylphenidate (MPH) and once with placebo. All medications will be administered orally with a capsule. The treatment order will be established by counterbalancing.

ELIGIBILITY:
Inclusion Criteria:

* The participant has been diagnosed with Mild Cognitive Impairment, either of the amnestic or the non-amnestic type.
* In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant signs and dates a written informed consent form.
* The volunteer is male or female.
* The participant is aged 60 to 80 years, inclusive, at the time of informed consent.
* The participant has a body mass index of 18.5-30, inclusive, at medical screening.
* The volunteer is healthy, i.e. absence of all exclusion criteria and has normal static binocular acuity (corrected or uncorrected) as well as normal hearing (using a whisper test during medical screening).

Exclusion Criteria:

* The subject has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may impact the ability of the subject to participate or potentially confound the study results.
* The volunteer has uncontrolled existing major psychiatric symptoms.
* The subject has uncontrolled hypertension.
* The volunteer has hyperthyroidism.
* The participant has known hypersensitivity to any component of the formulation of MPH or related compounds.
* The participant has glaucoma.
* The subject has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the first visit or is unwilling to agree to abstrain from alcohol from 24 hours prior to each test day and/or drugs throughout the study.
* The participant has any sensory or motor deficits which could reasonably be expected to affect test performance.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Verbal Learning Test Immediate Recall | 140 min after drug intake
Verbal Learning Test Delayed Recall | 175 min after drug intake
Verbal Learning Test Recognition | 180 min after drug intake
  Accuracy and reaction time
Amplitude of the N400 and P600 event-related potential (ERP) components | 140-190 min after drug intake
  during encoding and recognition of words of VLT, measured with EEG

SECONDARY OUTCOMES:
Performance on visual and auditory N-back test | 150 minutes after drug intake
Performance on a sustained attention to response task (SART) | 165 minutes after drug intake
Performance on a motor task | 170 minutes after drug intake
Amplitude of ERP components during the visual and auditory N-back test | 150-165 minutes after drug intake
Amplitude of ERP components during SART | 165 - 170 minutes after drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Anke Sambeth, Dr., Principal Investigator — Maastricht University
Locations (1):
- Orbis Medical Centre, Sittard-Geleen, Limburg, Netherlands